CLINICAL TRIAL: NCT07114900
Title: Developing a Tailored, Theoretically-Driven Smartphone Physical Activity Intervention for African American Women: RCT
Brief Title: Randomized Controlled Physical Activity App Intervention for Black Women
Acronym: PA4HealthRCT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Marie Aline Sillice, PHD, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA4Health RCT; K23MD014164 (NIH); RB2023-00444 (Other: Institutional Review Board, Stony Brook University)
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Physical Activity
Keywords: Physical activity app, Wellness Text messaging, RCT
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: PA4Health app physical activity intervention (Experimental): The arm for the PA4health app intervention consists of six components: 1) Goal setting and monitoring, 2) Tailored motivational messages based on survey data on barriers and facilitators of physical activity, 3) Education, which consists of twenty-two physical activity (PA) related topics, 4) a semi-structured chatroom where 3-5 participants per chatroom interact with one another to receive and provide peer support for PA, 5) Locator, which provides information about community resources (e.g., community parks, museums) based on participant's zip code, and 6) Steps, which allow participant to monitor their daily level of exercise. Participants wear a Fitbit tracker during the program Edit
  Interventions: Behavioral: PA4Health app physical activity intervention
- Wellness Text Messaging (Active Comparator): Participants set goal for PA and are encouraged to monitor their level of physical throughout the program. They receive a daily wellness related message during the program as a contact control. They also wear Fitbit tracker during the program.
  Interventions: Behavioral: Wellness Text Messaging Program

INTERVENTIONS:
Behavioral: PA4Health app physical activity intervention — PA4Health app intervention Arm Description: During the app intervention consists of six components: 1) Goal setting and monitoring, 2) Tailored motivational messages based on survey data on barriers and facilitators of physical activity, 3) Education, which consists of twenty-two physical activity (PA) related topics, 4) a semi-structured chatroom where 3-5 participants per chatroom interact with one another to receive and provide peer support for PA, 5) Locator, which provides information about community resources (e.g., community parks, museums) based on participant's zip code, and 6) Steps, which allow participant to monitor their daily level of exercise. Participants wear a Fitbit tracker during the program
  Other Names: Behavioral PA4Health app physical activity intervention; PA4Health
  Arms: Behavioral: PA4Health app physical activity intervention
Behavioral: Wellness Text Messaging Program — Participants set goal for PA and are encouraged to monitor their level of physical throughout the program. They receive a daily wellness related message during the program as a contact control. They also wear Fitbit tracker during the program.
  Arms: Wellness Text Messaging

SUMMARY:
The goal of this study is test whether a physical activity app intervention compared to wellness text messaging intervention is more acceptable/engaging among Black women who want to increase their level of physical activity.

DETAILED DESCRIPTION:
The goal of this K23 aim is to examine the acceptability and feasibility of the 8-week PA4Health intervention compared to a general wellness text program with 3 assessments (baseline, post-intervention [8 weeks] and 6 months). Participants will complete a single counseling session prior to starting the program. They complete an objective measure of physical activity by wearing an accelerometer for one week at each assessment time point. During the intervention, they will provided with a Fitbit wrist tracker, that will be synchronized to the app, to be worn during the 8-week intervention. Participants will be able to set goals for physical activity as well as monitor their progress toward achieving their goals. Following the trial, they will complete self-reports survey as well as objective measures of physical activity. They will also complete a single qualitative interview to assess their experience with the intervention and to provide feedback for modification.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were:

* ages 18-64,
* Identify as AA and female
* own a smartphone
* be able to provide consent
* not regularly physically active (i.e. less than 90 mins. of MVPA per week,
* medically cleared for PA
* have a valid email address, and 9) no previous engagement in the study.

Exclusion Criteria:

individuals were excluded if they report

. physical limitations to PA engagement

* significant medical conditions (e.g. heart failure)
* planned surgery in the next 6 months
* pregnant or plan to become pregnant in the next 6 months

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants identified as female or woman
Enrollment: 50 (Actual)
Dates: Start 2025-03-09 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS)--app satisfaction | End of 8 weeks
  Description: The SUS measures ability of technology software. High levels of usability and acceptability of the app will be determined by a score greater than 70 on the SUS. Information will be used for improvement of the software.
  Time Frame: 8 weeks study
Metada data collected from app system | 8 weeks
  This information will inform usage of patterns of participants, including how frequently the logged into the app system and the component of the app the more frequently or less frequently Time Frame: 8weeks

SECONDARY OUTCOMES:
Accelerometer/actigraph data | baseline, 8 weeks, 6-month follow-up
  Actigraph data will be analyzed to explore potential changes over time objectively collected min/week of MVPA
Physical activity constructs | baseline, 8 weeks, 6-month follow-up
  Assess changes in theoretical related constructs for physical activity, Stages of Change, Self-efficacy for Exercise, Physical Activity Enjoyment. Changes in mean scores from baseline to end intervention (8 weeks) will be assessed. Additionally changes in mean scores for these measures from end of intervention (8 weeks) and 6 month follow-up after controlling for baseline will be be explored.
Fitbit data | Participants will wear this device daily during the active phase of the 8-week intervention and also until follow-up/ 6-month follow up
  Fitbit data will be explored to estimate the effect of the intervention on mean steps/week over time

CONTACTS AND LOCATIONS:
Overall Officials: Marie Aline Sillice, PHD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
This was not part of the study protocol or informed consent. However, we will consider request to provide that information on an individual basis